CLINICAL TRIAL: NCT04077866
Title: B7-H3-Targeted Chimeric Antigen Receptor (CAR) T Cells in Treating Patients With Recurrent or Refractory Glioblastoma
Brief Title: B7-H3 CAR-T for Recurrent or Refractory Glioblastoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo Yinzhou People's Hospital (Unknown); Huizhou Municipal Central Hospital (Other); BoYuan RunSheng Pharma (Hangzhou) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU-RCT-BP102
Record Dates: First submitted 2019-08-26; First posted 2019-09-04 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Recurrent Glioblastoma; Refractory Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temozolomide alone (Active Comparator): Temozolomide will be given to patients orally every 5 days with 23 days interval. The initial dose is 150 mg/m2 on the first day and 200 mg/m2 for the rest if no toxicity is seen. If 200 mg/m2 is toxic, the drug will return to 150 mg/m2 or will be stopped.
  Interventions: Drug: Temozolomide
- Temozolomide + B7-H3 CAR-T (Experimental): Temozolomide will be given to patients orally every 5 days with 23 days interval. The initial dose is 150 mg/m2 on the first day and 200 mg/m2 for the rest if no toxicity is seen. If 200 mg/m2 is toxic, the drug will return to 150 mg/m2 or will be stopped.
  The B7-H3 CAR-T will be administrated via intratumoral or Intracerebroventricular injection through an Ommaya catheter in between Temozolomide cycles. Temozolomide treatment in the cycles of B7-H3 CAR-T treatment will be stopped.
  Interventions: Drug: Temozolomide; Biological: B7-H3 CAR-T

INTERVENTIONS:
Drug: Temozolomide — Temozolomide is an FDA-approved drug that is given to patients
  Other Names: TMZ
Biological: B7-H3 CAR-T — B7-H3-targeting CAR-T cells derived from patient own peripheral blood mononuclear cells will be given to patients via intracerebral injection though an Ommaya catheter
  Arms: Temozolomide + B7-H3 CAR-T

SUMMARY:
This is a randomized, parallel-arm, phase I/II study to evaluate the safety and efficacy of B7-H3 CAR-T in between Temozolomide cycles comparing to Temozolomide alone in treating patients with glioblastoma that has come back or does not respond to the standard treatment. The antigen B7-H3 is highly expressed in glioblastoma of a subset of patients. B7-H3 CAR-T, made from isolated patient peripheral blood mononuclear cells, can specifically attack patient glioblastoma cells that expressing B7-H3.

DETAILED DESCRIPTION:
Background

* B7-H3 is expressed in 70% of patients with glioblastoma
* B7-H3 is not expressed in normal tissues especially not in central nervous system. Therefore, it is an attractive GBM target for CAR-T therapy
* The investigators constructed a retroviral vector encoding a chimeric antigen receptor (CAR) targeting B7-H3, which can mediate CAR transfer into patient T cells with high efficiency.

Objectives

* To evaluate the safety and tolerability intratumoral/intracerebroventricular injection of B7-H3 CAR-T when used in between Temozolomide cycles
* To compare the overall survival (OS) and progression-free survival (PFS) of R/R GBM patients treated with B7-H3 CAR-T in between Temozolomide cycles vs Temozolomide alone
* To access the pharmacokinetics and pharmacodynamics of B7-H3 CAR-T in between Temozolomide cycles

Design

* Experimental group: Patients autologous T cells are activated and transduced with retrovirus containing B7-H3 CAR. CAR-T cells are expanded ex vivo and infused back to patients via intratumoral or intracerebroventricular injection through an Ommaya catheter. 3 injections of CAR-T are planned at two different doses with 1-2 weeks intervals. The CAR-T injections occur in between Temozolomide (TMZ) cycles. Temozolomide treatment during the cycles of CAR-T injections will be stopped and resumed next cycle. Patients may receive additional CAR-T cycles at the discretion of the principal investigator and oncologist.
* Control group: Patients will receive regular cycles of Temozolomide treatment with 5 days of treatment and 23 days of interval.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.
* Histologically confirmed diagnosis of World Health Organization (WHO) classification grade IV glioblastoma (GBM).
* Clinical Pathology confirms B7-H3 positive tumor expression by immunohistochemistry (IHC) at the initial tumor presentation or recurrent disease (H-score >= 50).
* Relapsed/refractory disease confirmed by radiographic evidence after standard therapy.
* Suitable for the surgery of the placement of the Ommaya catheter.
* Eastern Cooperative Oncology Group (ECOG) =0 or 1 (need to be confirmed before intratumoral or intracerebroventricular injection)
* >= 8 weeks after completion of front-line radiation therapy
* >= 6 weeks after completion of nitrourea chemotherapy
* >= 14 days after completion of Temozolomide or other chemotherapy
* 2 weeks of wash-out time after completion of targeted therapy with related adverse events (AE) on baseline (4 weeks for Bevacizumab). Patients with other chronic AEs are in the investigator's judgement
* Blood cell count： White blood count (WBC) >= 2000/μL；Neutrophil count >= 1500/μL；Platelets >= 100 x 103/μL；Hemoglobin >= 9.0 g/dL
* Serum Creatinine <= 1.5×ULN or Creatinine Clearance Rate (Cockcroft and Gault) > 30 mL/min/1.73 m2
* Alanine Transaminase (ALT) <= 5×ULN and total bilirubin < 2.0mg/dL
* Lung function: Oxygen (O2) saturation >= 92% on room air and < CTCAE grade 1 dyspnea
* Heart function: Left ventricular ejection fraction (LVEF) >= 40% by multigated acquisition (MUGA) scan or echocardiogram
* Normal coagulation function: prothrombin time (PT)，activated partial thromboplastin time (APTT) and international normalized ratio (INR)
* Good blood vessel condition for leukapheresis
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity within one year after B7-H3 CAR-T infusion

Exclusion Criteria:

* Other active malignancy in the past 2 years except non-melanoma skin cancer, completely surgical removed low grade tumor, post-therapeutic limited-stage prostate cancer, biopsy confirmed in situ cervical carcinoma, PAP test confirmed squamous intraepithelial lesions
* Participant is undergoing or planning to take other anti-tumor therapies
* Participant is systematic steroid-dependent, or is expecting to be treated with systematic steroid
* Active immunodeficiency virus (HIV) or hepatitis B or hepatitis C virus infection
* Active infection from fungi, bacteria and/or viruses
* Known history of the following cardiac diseases in the past 6 months: New York Heart Association (NYHA) defined grade III or IV heart failure, cardiac angioplasty, myocardial infarction, unstable angina and other clinically significant heart diseases
* Known history and/or clinically evident central nerve system diseases: seizure, epileptic seizure, aphasia, paralysis, stroke, severe brain damage, dementia, Parkinson's Disease, cerebellar diseases, organic brain syndrome and psychiatric disorders
* Autoimmune diseases
* Pregnant or breastfeeding females
* Therapeutic doses of corticosteroid within 7 days before leukapheresis or 72 hours before B7-H3 CAR-T infusion
* Cytotoxic chemotherapy without lymphocytotoxicity within 1 week before leukapheresis except that the treatment has been stopped for more than 3 half-lives of the drug
* Lymphocytotoxic chemotherapy (cyclophosphamide, Ifosfamide and bendamustine) within 2 weeks before leukapheresis
* Other clinical trials drugs within 4 weeks before leukapheresis except that the drug has no effect or the disease has progressed, and the treatment has been stopped for more than 3 half-lives of the drug
* Radiotherapy within 6 weeks before leukapheresis
* Prior trials of CAR-T or other cell therapy
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years, up to 15 years if necessary
  Kaplan Meier methods will be used to estimate median OS

SECONDARY OUTCOMES:
Incidence and type of adverse events | 12 weeks
  Number of Participants With Treatment-Related Adverse Events and Types of adverse events as Assessed by CTCAE v4.0
Maximum tolerated dose (MTD) | 12 weeks
  The highest dose of B7-H3 CAR-T that does not cause targeted dose-limiting toxicity
Progression-free survival (PFS) | 2 years, up to 15 years if necessary
  Kaplan Meier methods will be used to estimate median PFS. Progression is defined by Response Assessment in Neuro-Oncology (RANO) criteria
Peak Concentration (Cmax) of B7-H3 CAR-T | 12 weeks
  Peak Concentration (Cmax) of B7-H3 CAR-T in peripheral blood (PB) and cerebral spinal fluid (CSF)
Area under the concentration versus time curve (AUC) of B7-H3 CAR-T | 12 weeks
  Area under the concentration versus time curve (AUC) of B7-H3 CAR-T in peripheral blood (PB) and cerebral spinal fluid (CSF)
Disease response (ORR, CR, PR, DOR) | 2 years, up to 15 years if necessary
  Objective Response Rate (ORR) will be assessed by comparison with baseline magnetic resonance imaging by RANO. Complete Response (CR) is disappearance of all measurable and non-measurable disease for at least 4 weeks. Partial Response (PR) is >/= 50% decrease in lesions for at least 4 weeks. Duration of Response (DOR) is the time between the initial response to the treatment and subsequent disease progression.

OTHER OUTCOMES:
Cytokine levels in PB and CSF | 12 weeks
  The concentration of cytokines (IL-1, IL-2, IL-6, IL-10, TNF-α, IFN-γ) in PB and CSF
T cell levels and phenotype | 12 weeks
  The chimeric antigen receptor (CAR) T and endogenous T cell levels and memory/effector phenotype detected in peripheral blood (PB), and cerebral spinal fluid (CSF) (absolute number per ul). Statistical and graphical methods will be used to describe persistence and expansion

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Ningbo Yinzhou People's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golubovskaya V. CAR-T Cells Targeting Immune Checkpoint Pathway Players. Front Biosci (Landmark Ed). 2022 Apr 2;27(4):121. doi: 10.31083/j.fbl2704121. PMID 35468680